CLINICAL TRIAL: NCT00938249
Title: Effects of Monascus Garlic Fermented Extract on Serum Triglyceride Level: a Double-Blind, Randomized Controlled Trial
Brief Title: Effects of Monascus Garlic Fermented Extract on Serum Triglyceride Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: Wakunaga Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Hiroshima University ( Fumiko Higashikawa )
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: eki-146
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Hypertriglyceridemias
Keywords: Moderately Elevated Serum Triglyceride
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Monascus Garlic Fermented Extract (Experimental)
  Interventions: Dietary Supplement: Monascus Garlic Fermented Extract
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Monascus Garlic Fermented Extract
  Arms: Monascus Garlic Fermented Extract
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the effect of monascus garlic fermented extract on serum lipid concentrations in subjects with moderately elevated serum triglyceride.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as based on medical history and physical examination
* Fasting serum triglyceride 120 to 200mg/dl
* Willing not to serve as blood donor during the study
* Informed consent signed

Exclusion Criteria:

* Female subjects who are pregnant or nursing a child
* Participation in any clinical trial up to 90 days before Day 1 of this study
* Renal or hepatic dysfunction
* Heart disease
* Under medication
* Subjects who are taking functional food designed for weight loss or serum lipid reduction

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Fasting triglyceride level | Every 4 weeks (Overall 20 weeks)

SECONDARY OUTCOMES:
Abdominal circumference | Every 4 weeks (Overall 20 weeks)
Visceral fat area by CT scan | Week 0 and Week 12
Serum total cholesterol and LDL cholesterol levels | Every 4 weeks (Overall 20 weeks)
Serum adiponectin level | Week 0 and Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Hiroshima University, Hiroshima, Hiroshima, Japan

REFERENCES:
- [Derived] Higashikawa F, Noda M, Awaya T, Ushijima M, Sugiyama M. Reduction of serum lipids by the intake of the extract of garlic fermented with Monascus pilosus: a randomized, double-blind, placebo-controlled clinical trial. Clin Nutr. 2012 Apr;31(2):261-6. doi: 10.1016/j.clnu.2011.10.008. Epub 2011 Oct 29. PMID 22041543